CLINICAL TRIAL: NCT00129415
Title: The Effectiveness of UVA1 and UVB Irradiation in the Treatment of Inflammatory Dermatoses: An Open Pilot Study
Brief Title: Ultraviolet (UVA and UVB) Light Therapy in the Treatment of Inflammatory Skin Conditions
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Yolanda Rosi Helfrich, Assistant Professor of Dermatology, Medical School, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Derm 446
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Atopic Dermatitis; Psoriasis; Alopecia; Mycosis Fungoides; Urticaria; Dermatoses; Stretch Marks
Keywords: UVA1; UVB; atopic dermatitis; psoriasis; alopecia; mycosis fungoides (CTCL); urticaria; inflammatory dermatoses; stretch marks
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis; Alopecia; Mycosis Fungoides; Urticaria; Skin Diseases; Striae Distensae; Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- UVA1 Irradiation (Experimental): UVA 1 Irradiation (Sellemed UVA1 light source) up to 130 J/cm2
  Interventions: Procedure: UVA1 Irradiation
- UVB Irridiation (Experimental): UVB Irradiation maximum dose of 4000 mJ/cm2
  Interventions: Procedure: UVB Irradiation

INTERVENTIONS:
Procedure: UVA1 Irradiation — The affected areas on the body will be treated with UVA1 (Sellemed UVA1 light source) for up to 5 times per week for 16 weeks. The UVA1 dose will be up to 130 J/cm2.
  Arms: UVA1 Irradiation
Procedure: UVB Irradiation — The affected areas on the body will be treated with UVB light for up to 5 times per week for 16 weeks. The maximum UVB dose will be 4000 mJ/cm2.
  Arms: UVB Irridiation

SUMMARY:
The purpose of this investigation is to study the effectiveness of longer wavelength UVA1 (340-400nm) or shorter wavelength ultraviolet B [UVB] (290-320nm) irradiation in the treatment of inflammatory skin conditions (such as: atopic dermatitis, psoriasis, mycosis fungoides, alopecia areata, stretch marks and urticaria).

This research study aims to evaluate the effectiveness of an investigational device which is similar in appearance to a "tanning bed" but which emits ultraviolet irradiation of a specific wavelength known as UVA1. This device has not been approved by the Food and Drug Administration (FDA) for general use in this country, as of yet, but it has been used quite successfully in Europe for several years in treating such conditions as scleroderma, atopic dermatitis, urticaria pigmentosa and other skin conditions.

Instead of UVA1 therapy, patients may receive ultraviolet radiation of a specific wavelength known as UVB. UVA1 light is a longer wavelength and therefore a lower energy wavelength than UVB. UVB light is often the light associated with getting a sunburn since it has a higher level of energy. UVB light has been used successfully in the treatment of many skin conditions.

DETAILED DESCRIPTION:
The purpose of this investigation is to study the effectiveness of longer wavelength UVA1 (340-400nm) or shorter wavelength UVB (290-320nm) irradiation in the treatment of inflammatory skin conditions. Inflammatory dermatoses refer to conditions like atopic dermatitis (eczema) and psoriasis in which circulating leukocytes (T cells, neutrophils, and monocytes) infiltrate the skin. The infiltrating cells may be of malignant phenotype as in mycosis fungoides (cutaneous T cell lymphoma-CTCL). Up to 50 patients with one of these diagnoses or related conditions will participate in this study. The affected areas on the body will be treated with UVA1 or UVB for up to 5 times per week for 16 weeks. The UVA1 dose will be up to 130 J/cm2. The maximum UVB dose will be 4000 mJ/cm2. This UVA1 dosing schedule has been safely used in Germany for treating patients with atopic dermatitis, mycosis fungoides, granuloma annulare, scleroderma, and urticaria pigmentosa. Subjects will be evaluated clinically at baseline, weeks 1, 2, 4, and then at monthly intervals. More frequent evaluation may be required depending on the condition being studied. Paired skin biopsies may be taken from involved and uninvolved (or treated and untreated) areas before and during UV therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 10-80 years
* Clinical diagnosis of inflammatory dermatoses such as atopic dermatitis, psoriasis, mycosis fungoides, alopecia areata, and urticaria.
* No disease states or physical conditions that would impair evaluation of the test site.
* Willing and able to receive UVA1 or UVB, as directed in the protocol; make evaluation visits; and follow protocol restrictions.
* Signed, written, witnessed, informed consent form.
* Must live within a reasonable driving distance of Ann Arbor, Michigan, and/or be able to attend all of the scheduled appointments during the study.

Exclusion Criteria:

* History of photosensitivity (development of hives or bumps with exposure to light).
* UVA1 or UVB irradiation hypersensitivity in a UVA1/UVB photo-provocation test.
* Pregnant or nursing women.
* Involved in an investigational study within the previous 4 weeks.
* Presence of bacterial superinfection.
* Taken oral therapy for skin condition within the last 4 weeks
* Topical steroid therapy within the last 2 weeks
* History of excessive scar formation or keloids

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2000-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Clinical assessment to determine the effectiveness of light treatment for skin condition | Subjects will be evaluated at weeks 1, 2, and 4, then every month until the end of the study

SECONDARY OUTCOMES:
Assays to be performed on biopsy specimens may include any or all of the following assays: in situ hybridization, immunohistologic analysis, in situ zymography, radioimmunoassay, and Western blot analysis | At completion of the study.
Photographs will also be taken. | Color photographs will be obtained at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: John J Voorhees, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Wang F, Garza LA, Cho S, Kafi R, Hammerberg C, Quan T, Hamilton T, Mayes M, Ratanatharathorn V, Voorhees JJ, Fisher GJ, Kang S. Effect of increased pigmentation on the antifibrotic response of human skin to UV-A1 phototherapy. Arch Dermatol. 2008 Jul;144(7):851-8. doi: 10.1001/archderm.144.7.851. PMID 18645136